CLINICAL TRIAL: NCT01313546
Title: A Comparison of Sartorius Vs. Quadriceps Evoked Motor Response for Femoral Nerve to Prevent Secondary Catheter Failure
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Dr. Imad Awad, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Sunnybrook_Women's
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Femoral nerve block; total knee arthroplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- quadriceps (Active Comparator): quadriceps muscular contraction
  Interventions: Other: Stimulation of quariceps muscle
- sartorius (Active Comparator): stimulation of sartorius muscle through femoral nerve
  Interventions: Other: Stimulation of quariceps muscle

INTERVENTIONS:
Other: Stimulation of quariceps muscle — stimulation of quadriceps muscle through the stimulating catheter
  Other Names: Medial stimulation; patellar twitches

SUMMARY:
Objective: Continuous nerve block (freezing the nerve) is needed for knee replacement surgery to reduce pain, increase rehabilitation and discharge patients home fast. A lot of time, money and hospital resources are invested in inserting these catheters. The aim of this study is to compare two end points used for insertion of continuous femoral nerve block and to see which one results in fewer failures on the surgical ward.

Methodology: Patients having total knee replacement surgery will be recruited in this study. Patients will be randomized into two groups. The continuous femoral nerve block catheter will be inserted using ultrasound and nerve stimulation with two different end points (certain muscle contraction).

Patients will be followed on day 1 and 2 after surgery to observe which catheter fails, how much pain the patient suffers and how much painkiller the patients used.

DETAILED DESCRIPTION:
Background:

Continuous femoral nerve block (c FNB) is a widely used regional anesthetic technique for many lower limb operations. It provides superior pain relief, faster ambulation, and shorter hospital stay and less risk of side effects when compared with patient controlled analgesia (PCA).

Stimulating catheters (SC): SC were introduced back in 1999 to provide an objective end point to guide the catheter position by maintaining the desired evoked muscle response.

Stimulating catheter for continuous femoral nerve block: Salinas et al compared stimulating catheters vs. non-stimulating catheter in volunteers having femoral nerve block. They maintained a quadriceps evoked muscle twitch < 0.5 mA through the stimulating catheter . They reported a block success of 100% via the stimulating catheters versus 85% via the non-stimulating catheters (P = 0.07) and a much dense motor block and pain scores with SC as compared to NSC.

Motor responses of the femoral nerve: With peripheral nerve stimulation of the femoral nerve, two responses may be elicited, sartorius muscle contraction (contraction of the sartorius muscle through stimulation of its muscular branch) or quadriceps muscle contraction or patella twitch (contraction of the quadriceps muscle through stimulation its respective muscular branches). The two divisions of the femoral nerve are in fact medial and lateral divisions rather than anterior and posterior . The medial division supplies the sartorius muscle and the lateral division supplies the quadriceps muscle and both divisions lay within close proximity in the same fascial plane. Several regional anesthesia texts states that the anterior branch, supplying a motor branch to sartorius is above the fascia iliaca and this is partly why this stimulation should not be sought for FNB because there would be inadequate spread around the femoral nerve. An anatomical study by Gustafson et al and other anatomical text have forfeited this theory , . Furthermore, the rectus femoris of quadriceps often gets part of its innervation from the same division supplying the sartorius muscle.

Most authors advocate preferentially searching the quadriceps muscle response as articular branches are derived from the posterior or lateral division of the femoral nerve . However, the success of femoral nerve block using either quadriceps or sartorius twitch has not been confirmed with randomised controlled trials.

Secondary catheter failure: is defined as the failure of the peripheral continuous nerve block to provide adequate pain relieve after the primary block was instituted. The incidence ranges from 10 - 40% depending on the definition used , , . A lot of time, money and hospital resources are invested in placing the peripheral nerve catheters with the objective of providing optimal pain management and faster recovery.

We hypothesized that the success of FNB using sartorius muscle twitch is equivalent to quadriceps muscle twitch response. To test this hypothesis, we will conduct a prospective randomized double-blind controlled trial comparing femoral nerve block at the inguinal crease using sartorius or quadriceps muscle twitch as an end point for stimulation via a stimulating catheter.

Methods:

With institutional ethical approval (Faculty of Medicine, University of Toronto, Canada) and having obtained written informed consent, we plan to recruit 40 patients, aged 18-75, ASA I-III scheduled to undergo unilateral total knee arthroplastly in this prospective, randomised, single blinded controlled trial.

Exclusion criteria: patients with a history of significant medical or psychiatric problems, BMI > 40, allergy to local anesthetic drugs, prior surgery in the inguinal region, neurological disease with sensory or motor deficit, and diabetic neuropathy.

In the block room: patients will be premedicated with acetaminophen 1000 mg, celecoxib 400 mg and gabapentin 400 to 600 mg as part of out multimodal pain regimen. After an 18-gauge IV cannula is placed, patients will receive midazolam (0.03 mg/kg) for anxiolysis and routine monitors will be attached.

Randomization: Patients will be randomized with random computer allocation into 2 groups: group 1 = sartorius muscle twitch (SMT), group 2 = quadriceps muscle twitch (QMT).

Continuous Femoral Nerve block: After aseptic skin disinfection and sterile draping of the inguinal region, a 38 mm broadband 13-6 MHz linear array ultrasound (US) probe (Philips HD 11XE, Bothell, WA) will be placed on the skin to locate the position of the femoral nerve at the inguinal crease. The ultrasound transducer will be covered with a sterile, transparent dressing TegadermTM HP (3M Heath Care, St. Paul, MN). Sterile conductivity gel Ultra/Phonic (Pharmaceutical Innovations TM, Newark, NJ) will be used. In plane or out of plane approach will be used to guide the tuohy needle towards the femoral nerve. A skin wheal will be raised with 2 to 3 mLs of local anesthetic solution (1% lidocaine), peripheral nerve stimulator (PNS) with an initial current output of 1mA (frequency 2Hz, pulse width 0.1ms) will be used to verify the type of evoked muscle response. The stimulating tuohy needle will be inserted at 45º angle to the skin, 1 cm lateral to the femoral artery pulsation towards the femoral nerve under ultrasound guidance. The anesthesiologist will seek either sartorius or quadriceps muscle evoked muscle response based on the random number allocation in sealed opaque envelopes. The stimulating needle will be adjusted and once the appropriate muscle twitch was obtained at a current of less than 0.4 mA, the catheter will be threaded 3-5 cm pass the needle tip while maintaining spread of local anesthetic solution in a short axis view. Plain ropivacaine 0.5% mixed with lidocaine 1% will be injected in increments of 5 mL after negative aspiration up to a total of 20 mL. To determine the spread of local anesthetic agent we divided the area around the femoral nerve into 8 pie-chart sectors with the femoral nerve in the middle. For documentation we will use a piece of transparency film with the pie chart of eight even sectors drawn on it . The film will be positioned over the US image such that the center of the pie chart is positioned on the middle of the femoral nerve and the upper edge of the film is parallel to the upper edge of the US image. Having done this, we could determine the local anesthetic spread and compare it between the two groups. Time to femoral nerve location (time needle entered the skin to localization of plexus with adequate twitch), time to catheter insertion (start to end of catheter insertion) and time to completion of drug injection (start to end of drug injection) will be documented.

Motor and Sensory assessment: Motor block of femoral nerve, and sensory block of the femoral, saphenous, and lateral femoral cutaneous nerves will be evaluated by a blinded observer every 5 minutes for a period of 30 minutes post block insertion. A 22 G hypodermic needle will used to assess sensation in the femoral nerve distribution: middle third medial thigh, lateral femoral cutaneous nerve: lateral thigh, and saphenous nerve: anteriomedial middle third leg . Sensation will be graded as 0 = normal sensation, 1 = dull sensation, and 2 = no sensation. Motor block evaluation was graded as 0 = full power, 1= partial block (paresis), 2 = complete block (paralysis). The quadriceps muscle strength will be assessed by grading the ability or inability to extend the leg of the operated limb against gravity after the hip is passively flexed at 45°. Complete femoral nerve block will be defined as complete loss of a sharp sensation at middle third medial thigh with complete inability to extend the knee joint after hip flexion at 45º after 30 minutes post block insertion.

After the completion of the 30 minutes assessment period, each patient will receive a sciatic nerve block and spinal anesthesia. Sciatic nerve block will be performed using the subgluteal approach with 20ml of 0.5% plain ropivicaine. Spinal anesthesia will be performed in the lateral position with the operated side uppermost. Intrathecal isobaric bupivacaine 10 mg with 10 µg of fentanyl will be injected under sterile conditions using 25 G whitacre needle.

Postoperative period: patients will receive acetaminophen 1000mg q6 hourly, celexocib 200mg q12 hourly and gabapentin 200mg q8 hourly given orally. Patients will also receive hydromorphone contin 3mg q8 hourly and a hydromorphone patient controlled analgesia (PCA) for breakthrough postoperative pain. Visual analogue scale (VAS) will be assessed 4 hourly for the first 48 hours. Total hydromorphone consumption and time of first PCA dose will be recorded. The patient will be given a 24 h diary to record VAS on. The research assistant will interview the patient on postoperative day one and two. VAS scores will be documented from the patient diary and the nursing records.

The primary end point of our study will be the number of secondary femoral nerve block failure 24 hours past catheter insertion. A dull needle will be used to test the sensory dermatomes for femoral nerve (mid thigh medial aspect). Normal sensation compared with the non-operative site will be considered as failure of the catheter. Secondary catheter failure is defined as the lack of impaired sensory deficit on the medial and anterior aspect of the mid thigh. The study is designed as a pilot study to obtain estimates upon which to base a future larger trial. As such a rigorous sample size calculation is not provided. The goal will be to recruit a minimum of 12 subjects per group, which is the number, required to construct a confidence interval (Statistical Rules of Thumb by Gerald van Belle, 2002, John Wiley and Sons). To account for potential drop out, the number will be increased to 20 per group.

Secondary outcomes include; time to perform the block, VAS scores at 24 hours, total oral hydromorphone use and hydromorphone PCA, and spread of local anesthetic around the femoral nerve. Statistical analysis will be performed using SAS Version 9.1 (SAS Institute, Cary, North Carolina, USA).

Implications:

* Operating room efficiency: an average femoral nerve catheter technique takes around 20-25 minutes to complete. Part of the delay in the execution of this procedure is eliciting quadriceps twitch through the stimulating catheter. If this study proves that the two elicited twitches as equally efficacious, it can shorten the procedure time by 7-10 minutes.
* Potential nerve injury: minimal tuohy needle manipulation could potentially reduce the risk of nerve injury
* Patient discomfort: Minimal needle manipulations will lead to decrease patient discomfort.

Referenc

ELIGIBILITY:
Inclusion Criteria:

* Patients having total knee arthroplasty AsA 1-3

Exclusion Criteria:

* patients with a history of significant medical or psychiatric problems, BMI > 40, allergy to local anesthetic drugs, prior surgery in the inguinal region, neurological disease with sensory or motor deficit, and diabetic neuropathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
the number of secondary catheter failures | 12 months
  to prevent the occurance of failed femoral nerve catheter on postoperative day 1

SECONDARY OUTCOMES:
total morphine consumption | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: imad Awad, FFARCSI, Principal Investigator — Sunnybrook Hospital
Locations (1):
- The Holland orthopedic and arthritic centre, Toronto, Ontario, Canada